CLINICAL TRIAL: NCT01584206
Title: Assessment of Sterol Metabolism in Sitosterolemia: A Pilot Study of Patients Treated With Ezetimibe
Brief Title: Sitosterolemia Metabolism
Acronym: STAIR7002
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B2011:051
Record Dates: First submitted 2012-04-16; First posted 2012-04-24 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2015-12

CONDITIONS: Sitosterolemia
Keywords: Sitosterolemia; Ezetimibe; Plant sterol; Cholesterol
MeSH Terms: conditions — Sitosterolemia | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ezetimibe (Experimental): Compare on and off ezetimibe
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — 10mg ezetimibe/day, at least 4 months

SUMMARY:
Ezetimibe has become the treatment choice for patients with sitosterolemia. Ezetimibe is an inhibitor of cholesterol absorption from the gastrointestinal tract. The purpose of this study is to determine if ezetimibe improves whole body plant sterol and cholesterol homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of homozygous sitosterolemia as established by genotyping and clinical parameters

Exclusion Criteria:

* pregnant
* intellectual disability
* major infectious diseases
* immunodeficiency
* cancer
* renal failure
* diabetes

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma cholesterol level | 8 months
  Plasma cholesterol level will be assessed by GC
Plasma sitosterol level | 8 months
  Plasma plant sterol assessment using GC

SECONDARY OUTCOMES:
Cholesterol absorption | 4 month
  Use stable isotope technique to assess cholesterol absorption
Cholesterol synthesis | 4 months
  Use of stable isotope to assess cholesterol synthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Semone B Myrie, PhD, Principal Investigator — University of Manitoba; Peter J Jones, PhD, Study Chair — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Othman RA, Myrie SB, Mymin D, Roullet JB, DeBarber AE, Steiner RD, Jones PJH. Thyroid Hormone Status in Sitosterolemia Is Modified by Ezetimibe. J Pediatr. 2017 Sep;188:198-204.e1. doi: 10.1016/j.jpeds.2017.05.049. Epub 2017 Jun 16. PMID 28625503
- [Derived] Othman RA, Myrie SB, Mymin D, Merkens LS, Roullet JB, Steiner RD, Jones PJ. Ezetimibe reduces plant sterol accumulation and favorably increases platelet count in sitosterolemia. J Pediatr. 2015 Jan;166(1):125-31. doi: 10.1016/j.jpeds.2014.08.069. Epub 2014 Oct 16. PMID 25444527